CLINICAL TRIAL: NCT04831242
Title: Monitoring Key Activity and Physiology of Neonates in Intensive Care
Acronym: Meerkat
Status: Recruiting | Type: Observational
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Kathryn Beardsall, Principle Investigator, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: Meerkat vs 1.0 1st Feb 2021
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Neonatal Seizure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To optimise and evaluate a novel non-contact physiological monitoring system in the neonatal intensive care unit (NICU)

DETAILED DESCRIPTION:
To optimise and evaluate a novel non-contact physiological monitoring system in the neonatal intensive care unit (NICU)

ELIGIBILITY:
Inclusion Criteria:

* written informed parental consent

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Newborn infants in neonatal intensive care
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Movement | First week of life
  cm

CONTACTS AND LOCATIONS:
Locations (1):
- Addenbrookes Hospital, Cambridge, United Kingdom